CLINICAL TRIAL: NCT03219359
Title: Maintenance in Autologous Stem Cell Transplant for Crohn's Disease (MASCT - CD)
Brief Title: Autologous Stem Cell Transplant for Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aaron Etra (Other)
Responsible Party: Sponsor-Investigator, Aaron Etra, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 17-0378
Record Dates: First submitted 2017-07-13; First posted 2017-07-17 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease
Keywords: IBD; Inflammatory Bowel Diseases; Gastroenteritis; Crohn's disease; Colitis; Vedolizumab
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases; Gastroenteritis; Colitis | interventions — Bone Marrow Transplantation; Cyclophosphamide; thymoglobulin; Methylprednisolone; vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Hematopoietic Stem Cell Transplant followed by maintenance Vedolizumab
  Interventions: Procedure: Autologous stem cell transplant; Drug: Cyclophosphamide; Drug: Thymoglobulin; Drug: Methylprednisolone; Drug: Vedolizumab

INTERVENTIONS:
Procedure: Autologous stem cell transplant — Hematopoietic stem cell transplantation
  Other Names: Bone Marrow Transplant
Drug: Cyclophosphamide — Days 1 and 2: Cyclophosphamide 2gm/m2/day x 2 days (total dose 4gm/m2) Day 3 until leukapheresis: G-CSF 10μg/kg/day to CD34+ >20x104/ml then leukapheresis daily to collection goal
Drug: Cyclophosphamide — Day -6 to -3: Cyclophosphamide 50 mg/kg/day (200 mg/kg total dose)
Drug: Thymoglobulin — Day -3 to -1: 2.5 mg/kg/day (7.5 mg/kg total dose)
  Other Names: ATG
Drug: Methylprednisolone — Day -3 to -1: 1 gram prior to each ATG dose
Drug: Vedolizumab — Starting first day after discharge from transplant admission, then 2 weeks after 1st infusion, 4 weeks after 2nd infusion, followed by every 8 weeks for 52 weeks (8 doses)

SUMMARY:
Crohn's Disease (CD) is an inflammatory bowel disease. It can lead to significant complications and discomfort in the stomach and intestines. Crohn's disease is a debilitating, incurable disease of immune cells; it affects almost 1 million people in the United States. CD is characterized by inflammation of the stomach and intestine as well as organs outside of the intestines such as the skin, eyes, and joints. Current therapies to treat CD aim to suppress the patient's immune cells but these therapies become ineffective for the majority of patients and lead to complications including the requirement for surgical bowel resection, impaired quality of life, and lifelong disability. Hematopoietic stem cell transplantation (HCT) is a procedure used to treat a number of medical conditions including Crohn's disease. To improve success of HCT in CD doctors considered combining transplant with other drugs to improve the chances of achieving remission and also maintaining the remission. The Investigators' plan in this study is to incorporate the drug Vedolizumab after transplant to test if this drug will improve remission and make patients healthier.

Patients may qualify to take part in this research study because Crohn's disease is active, because surgery is not a treatment option and because there is evidence that the disease has failed to respond to treatments for Crohn's disease including the following:

* corticosteroids
* azathioprine, 6-mercaptopurine, methotrexate
* Anti-TNFα (infliximab, adalimumab, certolizumab, golimumab)
* Anti-integrin agents (natalizumab, Vedolizumab) If patients meet entry criteria will undergo a baseline endoscopy, colonoscopy and MR or CT enterography. If documentation of active mucosal disease patients will then be tapered off of current medications and undergo stem cell mobilization. Mobilization will involve low dose chemotherapy, growth factors and require 1-2 week hospitalization. Patients will then undergo stem cell transplant which will involve high dose chemotherapy and require a 2-4 week hospitalization. After restoration of the immune system patients will be placed on vedolizumab per standard dosing (0,2,6 then 8 every weeks) for a total of 8 doses. Patients will have monthly study visits and a repeat colonoscopy and MR/CT scan at 6 months.

DETAILED DESCRIPTION:
Crohn's Disease Inflammatory bowel disease, encompassing Crohn's disease (CD) and ulcerative colitis (UC), represent incurable chronic inflammatory disorders of the intestinal tract. Patients with IBD experience a chronic relapsing and remitting course of their disease, with little ability to predict when these flares will occur. The primary symptoms of IBD are related to inflammation of the gastrointestinal (GI) tract and include diarrhea, hematochezia, and abdominal pain. Patients also frequently suffer from systemic inflammatory symptoms such as fatigue, arthritis, uveitis, and erythema nodosum.

Current therapies for CD are directed at symptom control by suppressing the immune system or surgical resection of the damaged bowel. The most efficacious medical therapy, the combination of an anti-tumor necrosis factor alpha (anti-TNFα) monoclonal antibody and an immunomodulator (6-MP or azathioprine), results in a 56% clinical remission rate at 6 months, leaving a large portion of patients with active disease. Unfortunately, even among initial responders to this therapy a large proportion of responders eventually relapse, requiring that the majority of patients with Crohn's disease ultimately need new therapeutic modalities.

The most promising treatment for CD patients refractory to anti-TNFα therapy, are inhibitors of T-cell trafficking to the GI tract. The first of these, natalizumab, was approved by the FDA in 2008 and is indicated for CD and multiple sclerosis. Natalizumab binds to the α4 integrins (α4β1 and α4β7), disrupting interaction with its ligands VCAM-1 and MAdCAM-1 and impeding leukocyte adhesion and trafficking to the CNS and GI tract respectively. The ENACT study demonstrated a 6% improvement in clinical response in patients receiving natalizumab compared to placebo (56% vs 49%, p = 0.05) in 905 patients with moderate to severe Crohn's disease defined as a CDAI score of between 220-450. While the overall therapeutic efficacy was modest, in a subgroup analysis of patients refractory to anti-TNFα therapy 55% of patients in the treatment arm responded compared to 35% in the placebo arm (P < 0.05). One negative feature of natalizumab is that general blockade of α4 integrins inhibits T-cell trafficking to the CNS in addition to the intestine and has been shown to increase the risk of progressive multifocal leukoencephalopathy (PML), a fatal infection caused by the JC Virus (JCV).

A newer monoclonal antibody, vedolizumab, binds only to α4β7 which results in selective inhibition of leukocyte trafficking to the intestine and theoretically eliminates the risk of PML. Vedolizumab was approved by the FDA in 2014 based on a randomized controlled trial of 368 patients with refractory CD treated with vedolizumab which demonstrated a significant induction of clinical remission in this cohort (14.5% vs 6.8%, p=0.02) . Similar to natalizumab, a subgroup analysis demonstrated that 10.5% of patients refractory to anti-TNFα therapies will respond to vedolizumab. Among vedolizumab responders who were randomized to maintenance vedolizumab, responders were more likely to be in clinical remission at week 52 compared to patients not on maintenance therapy (39% vs 22%, p=0.001).

Autologous hematopoietic stem cell transplantation (HCT) is a procedure used to treat and/or cure a number of malignant conditions including lymphoma and myeloma. Briefly, following collection and cryopreservation of hematopoietic stem cells, very high doses of chemotherapy to overcome tumor resistance are given followed by reinfusion of the collected hematopoietic stem cells. The transplanted HSC reconstitute the marrow and restore normal blood cell production and reconstitute the immune system. More recently, autologous HCT has been shown to be an effective treatment in a number of autoimmune disorders such as multiple sclerosis, scleroderma, and CD. For autoimmune disorders, the presumptive mechanism of action is that intensive immunoablation followed by reinfusion of hematopoietic cells results in an immunological "reset" without recurrence of the autoimmune disease. The most common chemotherapy regimen used for autoimmune disorders is a combination of cyclophosphamide with anti-thymocyte globulin. The safety of this regimen is well established and has been recommended for the previously mentioned conditions by the European Group for Blood and Marrow Transplantation (EBMT).

Stem cell transplantation for CD has been recognized as a potential therapeutic modality since the 1980s. Northwestern University treated 24 patients with CD where stem cells were mobilized with cyclophosphamide 2 mg/m2 and G-CSF 10 mcg/kg/day followed by an immunoablative transplant using cyclophosphamide 200 mg/kg (50 mg/kg daily for 4 days) and ATG (30 mg/kg) as per the previously referenced consensus statement by EBMT. In this study there was no treatment related mortality and clinical relapse-free survival (defined as not restarting CD therapy) was 73% (17/23) at 1 year but declined to 19% at 5 years demonstrating the problem of durable disease control with autologous transplant alone. Interestingly, 8/15 (53%) patients who restarted therapy for recurrent Crohn's symptoms were able to achieve clinical remission, highlighting the possibility that efficacy of medications previously used can be restored following autologous HSCT. Autologous Stem-Cell Transplantation in Crohn's Disease (ASTIC) trial randomized patients either to autologous transplantation or stem cell mobilization chemotherapy without transplantation. This trial design allowed for the benefit of autologous HCT to be assessed independently of the potential benefit of the immunosuppression from high dose cyclophosphamide used to mobilize stem cells. The primary endpoint of the trial was assessed by the Crohn's Disease Activity Index (CDAI), the most prevalent method of assessing Crohn's disease clinical activity, where a level <150 is considered to represent disease remission. The ASTIC trial demonstrated at 1 year in patients who underwent transplant 44% were in clinical remission compared to 9% of patients who underwent mobilization only (p = 0.017). One death occurred in this study believed secondary to cyclophosphamide induced sinusoidal obstructive syndrome. Across all studies there has been one treatment related death out of 69 transplanted patients (1%), which is approximately the rate expected with autologous HCT for a malignancy such as multiple myeloma and significantly lower than the 5-10% expected transplant related mortality for other malignancies like lymphoma. Additional support for the safety of autologous HCT for autoimmune disorders comes from similarly designed studies using the same conditioning regimen of cyclophosphamide and ATG for other autoimmune or connective tissue disorders. For example, the one year mortality rate following autologous transplantation in 129 relapsing-remitting multiple sclerosis patients was 0%.

The discrepancy in response rates between the ASTIC study (44%) and the Northwestern study (73%) are likely due to several factors. First, the Northwestern population included patients with less severe Crohn's disease than the ASTIC trial. The Northwestern patients were eligible provided that the patient failed anti-TNF therapy while the ASTIC trial used stricter eligibility criteria. In addition, the ASTIC trial required endoscopic evidence of active Crohn's disease and therefore excluded patients whose disease activity scores reflected causes other than active inflammatory Crohn's disease, while the Northwestern trial did not. The CDAI score can be inflated from symptoms related to functional bowel disease and not the active inflammatory disease which is the target of immunosuppressive therapies. Active inflammatory mucosal disease is the greatest predictor of disease free survival and improves the reliability of the CDAI as a disease activity index. Finally, in an unknown number of patients the primary endpoint for the Northwestern patients was assessed on the basis of telephone report from patients that were asymptomatic and not on immunosuppressants, rather than the more rigorous CDAI score.

Based on the successes described in transplanting Crohn's disease patients and guidelines on transplant utilization developed by the EBMT, other centers have begun to open their own transplant programs under the auspices of clinical trials.

High doses of cyclophosphamide (high-CY), at a dose of 50 mg/kg/day X 4 days has become a standard dosing regimen in transplantation, a standard dosing for other transplant studies in Crohn's Disease, and the chemotherapeutic agent proposed for this clinical trial's Crohn's disease conditioning regimen. In this study, high-CY will be combined with an additional immunosuppressant, rabbit anti-thymocyte globulin (thymoglobulin, ATG), which has become part of the autologous transplant approach for autoimmune diseases including Crohn's disease. Thymoglobulin is a rabbit-thymocyte globulin obtained from the serum of rabbits immunized with human thymus lymphocytes. ATG is a lymphocyte-selective immunosuppressant that acts by causing in vivo T-cell depletion in blood and lymphoid tissues . There are sustained shifts in T and B cell subpopulations from memory to naïve cell dominance, supportive of thymic reprocessing and reeducation of the reconstituting immune system. This, in essence, resets the immune system of patients with autoimmune diseases, of which Crohn's disease may be considered. Thymoglobulin, the brand of ATG being used in this study, has a half-life of 2-3 days. This allows for further delay in the return of activating T cells which contribute to the pathophysiology of Crohn's disease.

Rationale for Incorporating Vedolizumab to Maintenance post Autologous Transplantation: While the results of the ASTIC trial suggest autologous BMT for CD is an effective therapy, there is still room for improvement as sustained remission is achieved in only 44% of patients. The reasons for the failure of induction of remission and the lack of sustained response in a portion of patients are unknown, but presumably recapitulation of the autoimmune response after transplant plays an important role. Vedolizumab is appealing to test after autologous stem cell transplant as it targets inflammatory T cells destined for the intestine (expressing α4β7). These T cells would be expected to be present in the graft and their blockade may improve the induction of remission achieved by the graft and leave the majority of protective T cells in the graft available to the recipient's recovering immune system. The addition of vedolizumab not only has the potential to improve induction of remission from the transplant itself but, as an adjunct therapy post-transplant, it may also help to maintain remission in this patient cohort. The need to provide patients with maintenance therapy post inductive therapy is well established both for medical therapeutics as well as post-operatively and vedolizumab has been established as an effective maintenance agent. The restoration of response to previously failed medications observed in other studies suggests that patients who did not respond to vedolizumab previously may now respond post HCT. This study will test the hypothesis that vedolizumab maintenance therapy will improve outcomes at 1 year post-transplant by decreasing the portion of patients whose disease recurs and increasing the portion of patients for whom the transplant induces remission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease by standard criteria
* Active disease based on clinical symptoms, defined as CDAI >250. In patients with an ostomy, the number of liquid stools score in the CDAI will be replaced by the number of times that the ostomy bag is emptied daily.
* Active disease based on endoscopic evaluation, defined as SES-CD score > 3 in at least one bowel segment
* Failure to respond to (or intolerant/adverse reaction to or declines) a member of each of the class of drugs listed below:

  1. corticosteroids
  2. azathioprine,
  3. 6-mercaptopurine, methotrexate
  4. Anti-TNFα (infliximab, adalimumab, certolizumab, golimumab)
  5. Anti-integrin agents (natalizumab, vedolizumab)
  6. Ustekinumab
* Failure to respond refers to ongoing objective inflammation with symptoms and, as is traditional, is defined by the gastroenterologist evaluating the patient.
* No surgical therapeutic option secondary to risk of short bowel syndrome or patient refusal

Exclusion Criteria:

* History of significant toxicity to any medications used in trial (cyclophosphamide, thymoglobulin, vedolizumab)
* Pregnant or breastfeeding
* Age <18
* Karnofsky Performance Score <60
* Patients who have an uncontrolled infection (presumed or documented) despite appropriate therapy for at least one month
* Patients with symptomatic coronary artery disease or uncontrolled congestive heart failure.
* HIV infected
* Ejection fraction <30% or requiring supplemental continuous oxygen.
* DLCO <35% or requiring supplementary oxygen.
* Patients for whom an insufficient number of stem cells (<2 X 10^6/kg) have been collected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-22 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Crohn's Disease Activity Index (CDAI) | baseline and 1 year post transplant
  The proportion of patients in clinical remission, defined as a CDAI < 150, one year after autologous HCT from 45% to 65% as compared to baseline.

SECONDARY OUTCOMES:
Change in endoscopic activity indices | baseline and 1 year post transplant
  The change in endoscopic activity indices (SES CD) following autologous HCT and vedolizumab maintenance as compared to baseline.The maximal score for the SES-CD is 56. Each of 5 segments of intestine (rectum, colon - descending, colon - ascending, colon - transverse, ileum) is scored from 0-3 on four parameters - ulceration, extent of ulceration, extent of disease and stenosis. A maximal score of 45 is possible for the first three parameters and 11 for stenosis as a score of 3 implies a stricture that cannot be traversed prohibiting evaluation of later segments. An SES score of 0-2 would be defined as mucosal healing as the presence of a single ulcer in one bowel segment would necessitate a minimal score of 3. A decrease of SES of 50% from baseline is felt to represent an endoscopic response.

OTHER OUTCOMES:
Change in burden of intestinal disease | baseline and 1 year post transplant
  The change in overall burden of intestinal disease (Magnetic resonance enterography ((MRE)+SES-CD) following autologous HCT and vedolizumab maintenance as compared to baseline.
Change in Inflammatory Bowel Disease Questionnaire (IBDQ) | baseline and 1 year post transplant
  The change in quality of life indices as evaluated via the IBDQ following autologous HCT and vedolizumab maintenance as compared to baseline. An increase in the IBD-Q of 16-32 points is generally considered meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Etra, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Louis Cohen, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided